CLINICAL TRIAL: NCT01162122
Title: A Phase III, Randomized, Controlled, Observer-Blind, Multicenter Study to Evaluate the Safety and Immunogenicity and the Consistency of Three Consecutive Lots of a MF59C.1 Adjuvanted Trivalent Subunit Influenza Vaccine in Elderly Subjects Aged 65 Years and Older
Brief Title: Safety and Immunogenicity of MF59C.1 Adjuvanted Trivalent Subunit Influenza Vaccine in Elderly Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V70_27
Record Dates: First submitted 2010-07-13; First posted 2010-07-14 (Estimated); Results first posted 2014-06-12 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Influenza
Keywords: Elderly; Influenza; Immunogenicity; Safety; Adjuvant; Adjuvanted; Adjuvants; Vaccines
MeSH Terms: conditions — Influenza, Human | interventions — fluad vaccine; Influenza Vaccines

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- aTIV (Experimental): Subjects received one dose of MF59-adjuvanted trivalent subunit influenza vaccine (aTIV) from one of three consecutive lots (Lot 1, Lot 2 or Lot 3).
  Interventions: Biological: MF59 adjuvanted trivalent subunit influenza vaccine (aTIV)
- Licensed TIV (Experimental): Subjects received one dose of non-adjuvanted trivalent subunit influenza vaccine (TIV).
  Interventions: Biological: Non-adjuvanted trivalent subunit influenza vaccine (TIV)

INTERVENTIONS:
Biological: MF59 adjuvanted trivalent subunit influenza vaccine (aTIV) — one dose 0.5 mL administered IM in the deltoid muscle of (preferably) the non-dominant arm
  Other Names: Fluad
  Arms: aTIV
Biological: Non-adjuvanted trivalent subunit influenza vaccine (TIV) — one 0.5 mL dose administered IM in the deltoid muscle of (preferably) the non-dominant arm
  Other Names: Agriflu
  Arms: Licensed TIV

SUMMARY:
The present phase III study aims to evaluate the safety and immunogenicity of MF59-adjuvanted subunit seasonal influenza vaccine and to evaluate the consistency in the manufacturing process of three consecutive lots of MF59-adjuvanted subunit seasonal influenza vaccine with respect to immunogenicity in subjects aged 65 years and older. The active comparator non-adjuvanted seasonal influenza vaccine is approved for use in this age group in the United States and will be used to provide a comparative assessment for immunogenicity and safety.

ELIGIBILITY:
Inclusion Criteria:

Males and females subjects aged ≥65 years at day of vaccination who are willing and able to comply to study procedures.

Exclusion Criteria:

1. Individuals with behavioral or cognitive impairment or a psychiatric condition or with a history of any illness that,in the opinion of the investigator, would have interfered with the subject's ability to participate in the study.
2. Individuals who were not able to comprehend and/or follow all required study procedures for the whole period of the study.
3. Known or suspected impairment/alteration of immune function.
4. Individuals with a known bleeding diathesis.
5. History of Guillain-Barré syndrome.
6. Individuals with history of allergy to vaccine components and/or a history of any anaphylaxis, serious vaccine reactions or hypersensitivity to influenza viral proteins, egg proteins (including ovalbumin), polymyxin, neomycin, betapropiolactone, thimerosal/ sodium ethylmercurothiosalicylate/ mercury and nonylphenolethoxylate/ nonoxynol-9 (spermicide).
7. Receipt of another investigational agent within 30 days prior to enrollment in the study or before completion of the safety follow-up period in another study.
8. Individuals who had received any other vaccines within 2 weeks for inactivated vaccines or 4 weeks for live vaccines prior to enrollment in this study or who had planned to receive any vaccine within 3 weeks from the study vaccine.
9. Individuals who had received vaccination against seasonal influenza in the previous 6 months.
10. Individuals with oral temperature ≥38.0°C (≥100.4°F) on day of study vaccination.
11. Individuals with history of substance or alcohol abuse within the past 2 years.
12. Individuals providing consent who did not consent to the retention of their serum samples after study completion.
13. Elective surgery or hospitalization planned to occur during the treatment phase or during the follow-up phase that, according to the opinion of the investigator, might have poses additional risk to the subject.
14. Subjects from whom blood could not be drawn at visit 1.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 7109 (Actual)
Dates: Start 2010-08; Primary Completion 2011-08 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (38):
- United States (21):
  - 301, Tatum Highlands Medical Associates PLLC, 26224 N Tatum Blvd 15A, Phoenix, Arizona
  - 318 Avail Clinical Research, 860 Peachwood Drive, DeLand, Florida
  - 306 Westside Center for Clinical Research, 810 Lane Avenue South, Jacksonville, Florida
  - 328 Miami Research Associates, 6141 Sunset Drive, Miami, Florida
  - 320 Johnson County Clin-Trials, 15602 College Blvd, Lenexa, Kansas
  - 316 Heartland Research Associates LLC - Axtell Clinic - PA, 700 Medical Center Dr, Newton, Kansas
  - 310 Heartland Research Associates LLC, 3730 N Ridge Road Suite 600, Wichita, Kansas
  - 322 Heartland Research Associates Wichita, 1709 S. Rock Road, Wichita, Kansas
  - 314 Saint Louis Univ Med Div of Infectious Diseases Immunology, 1100 S Grand Blvd DRC- Rm 827, St Louis, Missouri
  - 330 Mercy Health Research, 12680 Olive Blvd Suite 200, St Louis, Missouri
  - 313 Clinical Research Center of Nevada, 7425 W Azure Suite 150, Las Vegas, Nevada
  - 311 Regional Clinical Research INC, 415 Hooper Road, Endwell, New York
  - 326 Triangle Medical Research, 5816 Creedmoor Rd. Suite 104, Raleigh, North Carolina
  - 332 Piedmont Medical Research, 1901 S. Hawthorne Rd. Suite 306, Winston-Salem, North Carolina
  - 303 Prestige Clinical Research, 333 Conover Drive, Franklin, Ohio
  - 325 Omega Medical Research, 400 Bald Hill Road, Warwick, Rhode Island
  - 312 Spartanburg Regional Medical Center, 485 Simuel Road, Spartanburg, South Carolina
  - 321 Jordan River Family Medicine, 1868 West 9800 South Ste 100, Jordan, Utah
  - 317 J. Lewis Research Inc., 2295 Foothill Drive, Salt Lake City, Utah
  - 305 Foothill Family Clinic South, 6360 South 3000 East, Salt Lake City, Utah
  - 323 PI Coor Clinical Research LCC, 10721 Main St Suite 1500, Fairfax, Virginia
- Colombia (4):
  - 209, Centro de Investigacion CAFAM, Avenida Carrera 68, Bogota D.C.
  - 206, Centro de Atencion e Investigacion Medica CAIMED, Carrera 42A, Bogota D.C.
  - 213, Centro de Atencion e Investigacion Medica CAIMED, Carrera 42A, Bogota D.C.
  - 207, Centro de Investigacion Cafesalud Medicina Prepagada, Cra 14 No Piso Sexto, Bogota D.C.
- Panama (2):
  - 203, Health Research International HRI, Clayton Ciudad Del Saber Edificio 118, Provincia de Panamá
  - 205, Medical and Research Center Calle 53 Urbanizacion Marbella, Consultorios Royal Center 108, Provincia de Panamá
- Philippines (11):
  - 103, De La Salle Health Sciences Institute, DBB B Dasmarinas, Cavite
  - 102, De La Salle Health Sciences Institute, Dbbb Dasmarinas, Cavite
  - 105, Manila Doctors Hospital, 667 United Nations Avenue, Ermita, Manila
  - 106, Our Lady of Lourdes Hospital, 46 P. Sanchez Street Sta., Mesa, Manila
  - 104 Jose Reyes Memorial Medical Center, Rizal Avenue Avenida Cruz, Manila
  - 107 Philippine General Hospital, Taft Avenue, Manila
  - 101, Asian Hospital and Medical Center 2205 Civic Drive Filinvest, Corporate City Alabang, Muntinlupa
  - 109, Research Institute for Tropical Medicine Department of Health Compound FILINVEST, Corporate City Alabang, Muntinlupa
  - 108, City Health Office 1 Rosa City, City Health Office 1, Rosa City
  - 110, San Juan de Dios Hospital, 2772 Roxas Blvd, Pasay
  - 111, St Lukes Medical Center, 279 E Rodriguez Sr Boulevard, Quezon City

REFERENCES:
- [Derived] Frey SE, Reyes MR, Reynales H, Bermal NN, Nicolay U, Narasimhan V, Forleo-Neto E, Arora AK. Comparison of the safety and immunogenicity of an MF59(R)-adjuvanted with a non-adjuvanted seasonal influenza vaccine in elderly subjects. Vaccine. 2014 Sep 3;32(39):5027-34. doi: 10.1016/j.vaccine.2014.07.013. Epub 2014 Jul 18. PMID 25045825

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from 4 sites in Columbia, 2 sites in Panama, 11 sites in Philippines, 21 sites in USA.
Pre-assignment Details: Five enrolled subjects were not randomized and did not receive study vaccination, hence were discontinued.
Groups:
- aTIV (Pooled): Subjects received one dose of MF59-adjuvanted trivalent subunit influenza vaccine (aTIV) from one of three consecutive lots (Lot 1, Lot 2 or Lot 3).
Period: Overall Study
Arm/Group | aTIV (Pooled) | Licensed TIV
Started | 3552 | 3552
Vaccinated | 3541 | 3541
Completed | 3361 | 3356
Not Completed | 191 | 196
Not completed — Withdrawal by Subject | 52 | 43
Not completed — Lost to Follow-up | 73 | 91
Not completed — Adverse Event | 3 | 2
Not completed — Death | 51 | 46
Not completed — Protocol Violation | 2 | 2
Not completed — Inappropriate enrollment | 5 | 4
Not completed — Administrative reason | 1 | 1
Not completed — Unable to classify | 3 | 7
Not completed — Missing primary reason | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline demography is described for safety set population.
  A vaccine different from the vaccine assigned at randomization was administered to 7 subjects in each vaccine group. For the safety analysis, these subjects were reassigned to the vaccine group for the vaccine they actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | aTIV (Pooled) | Licensed TIV | Total
Number analyzed (Participants) | 3545 | 3537 | 7082
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.0 (5.3) | 71.8 (5.3) | 71.9 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2272 | 2342 | 4614
  Male | 1273 | 1195 | 2468

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers in Subjects After Receiving One Dose of Lot 1 or Lot 2 or Lot 3 of aTIV
Description: Immunologic equivalence of 3 consecutive production lots of aTIV (Lot 1, Lot 2 and Lot 3), was assessed in terms of Hemagglutination Inhibition (HI) Geometric Mean Titers (GMTs) in subjects, at three weeks after vaccination, against each vaccine strain.
Time Frame: Day 22 post vaccination
Population: Analysis was done on the per protocol set population (PPS) i.e all randomised subjects who received the correct vaccine, provided evaluable serum samples, and had no major protocol deviation prior to unblinding.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- aTIV_Lot 1: Subjects received one dose of MF59-adjuvanted trivalent subunit influenza vaccine (aTIV) from Lot 1
- aTIV_Lot 2: Subjects received one dose of MF59-adjuvanted trivalent subunit influenza vaccine (aTIV) from Lot 2
- aTIV_Lot 3: Subjects received one dose of MF59-adjuvanted trivalent subunit influenza vaccine (aTIV) from Lot 3
Arm/Group | aTIV_Lot 1 | aTIV_Lot 2 | aTIV_Lot 3
Number analyzed (Participants) | 1073 | 1078 | 1076
Titers
  H1N1 strain (N=1072,1078,1075) | 209 [189 to 231] | 187 [170 to 207] | 199 [180 to 220]
  H3N2 strain (N=1072,1078,1075) | 548 [502 to 598] | 542 [498 to 591] | 556 [510 to 606]
  B strain | 56 [51 to 61] | 56 [51 to 61] | 58 [53 to 64]
Statistical Analysis 1: Comparison: aTIV_Lot 1 vs aTIV_Lot 2; Test type: Non-Inferiority or Equivalence — The 95% CIs of GMT ratios for the pairwise lot-to-lot group comparisons should fall within the equivalence range of 0.67 to 1.5; GMT ratio (H1N1 strain) = 1.12, 95% CI 2-sided [1 to 1.24]
Statistical Analysis 2: Comparison: aTIV_Lot 1 vs aTIV_Lot 3; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; GMT ratio (H1N1 strain) = 1.05, 95% CI 2-sided [0.95 to 1.17]
Statistical Analysis 3: Comparison: aTIV_Lot 2 vs aTIV_Lot 3; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; GMT ratio (H1N1 strain) = 0.94, 95% CI 2-sided [0.85 to 1.05]
Statistical Analysis 4: Comparison: aTIV_Lot 1 vs aTIV_Lot 2; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; GMT ratio (H3N2 strain) = 1.01, 95% CI 2-sided [0.92 to 1.11]
Statistical Analysis 5: Comparison: aTIV_Lot 1 vs aTIV_Lot 3; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; GMT ratio (H3N2 strain) = 0.99, 95% CI 2-sided [0.9 to 1.08]
Statistical Analysis 6: Comparison: aTIV_Lot 2 vs aTIV_Lot 3; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; GMT ratio (H3N2 strain) = 0.98, 95% CI 2-sided [0.89 to 1.07]
Statistical Analysis 7: Comparison: aTIV_Lot 1 vs aTIV_Lot 2; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; GMT ratio (B strain) = 1, 95% CI 2-sided [0.91 to 1.1]
Statistical Analysis 8: Comparison: aTIV_Lot 1 vs aTIV_Lot 3; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; GMT ratio (B strain) = 0.96, 95% CI 2-sided [0.87 to 1.05]
Statistical Analysis 9: Comparison: aTIV_Lot 2 vs aTIV_Lot 3; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; GMT ratio (B strain) = 0.96, 95% CI 2-sided [0.87 to 1.05]

2. Primary Outcome: Comparison of aTIV Versus TIV in Terms of Geometric Mean Titers (GMTs) Against Homologous Strains - PPS
Description: The non-inferiority of HI antibody responses of aTIV compared to TIV assessed in terms of post vaccination GMTs at three weeks after vaccination against the three homologous vaccine strains.
Time Frame: Day 22 post vaccination
Population: Analysis was done on PPS.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | aTIV (Pooled) | Licensed TIV
Number analyzed (Participants) | 3227 | 3259
Titers
  H1N1 strain (N=3225,3257) | 198 [185 to 211] | 141 [132 to 150]
  H3N2 strain (N=3225,3256) | 544 [513 to 575] | 337 [319 to 357]
  B strain | 55 [52 to 58] | 48 [46 to 51]
Statistical Analysis 1: Comparison: aTIV (Pooled) vs Licensed TIV; Test type: Non-Inferiority or Equivalence — Non-inferiority was established if the lower bound of the 95% CI for the day 22 vaccine group GMT ratios for all 3 homologous strains was >0.67; GMT ratio (H1N1 strain) = 1.4, 95% CI 2-sided [1.32 to 1.49]
Statistical Analysis 2: Comparison: aTIV (Pooled) vs Licensed TIV; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; GMT ratio (H3N2 strain) = 1.61, 95% CI 2-sided [1.52 to 1.7]
Statistical Analysis 3: Comparison: aTIV (Pooled) vs Licensed TIV; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; GMT ratio (B strain) = 1.15, 95% CI 2-sided [1.08 to 1.21]

3. Primary Outcome: Comparison of aTIV Versus TIV in Terms of Percentage of Subjects Achieving Seroconversion Against Homologous Strains-PPS
Description: The non-inferiority of HI antibody responses of aTIV compared to TIV assessed in terms of percentage of subjects achieving seroconversion at three weeks after vaccination against the three homologous vaccine strains.
  Seroconversion defined as prevaccination HI titer <10 and postvaccination HI titer ≥40 or at least a 4-fold increase in HI titers from prevaccination HI titer ≥10.
Time Frame: Day 22 post vaccination
Population: Analysis was done on PPS.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | aTIV (Pooled) | Licensed TIV
Number analyzed (Participants) | 3227 | 3259
Percentage of subjects
  H1N1 strain (N=3225,3257) | 77.4 [75.9 to 78.9] | 67.6 [65.9 to 69.2]
  H3N2 strain (N=3225,3256) | 74.0 [72.4 to 75.5] | 60.7 [59.0 to 62.3]
  B strain | 47.0 [45.2 to 48.7] | 41.2 [39.5 to 43.0]
Statistical Analysis 1: Comparison: aTIV (Pooled) vs Licensed TIV; Test type: Non-Inferiority or Equivalence — Non-inferiority was established if the lower bound of the 95% CI for the day 22 differences in seroconversion rates for all 3 homologous strains was ≥-10%; Group difference (H1N1 strain) = 9.2, 95% CI 2-sided [7.1 to 11.3]
Statistical Analysis 2: Comparison: aTIV (Pooled) vs Licensed TIV; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Group difference (H3N2 strain) = 12.7, 95% CI 2-sided [10.5 to 14.9]
Statistical Analysis 3: Comparison: aTIV (Pooled) vs Licensed TIV; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Group difference (B strain) = 5.2, 95% CI 2-sided [3.0 to 7.4]

4. Primary Outcome: Comparison of aTIV Versus TIV in Terms of GMTs Against Homologous Strains-Full Analysis Set (FAS)
Description: The superiority of HI antibody responses of aTIV compared to TIV assessed in terms of post vaccination GMTs at three weeks after vaccination against the three homologous vaccine strains.
Time Frame: Day 22 post vaccination
Population: Analysis was done on FAS i.e all randomized subjects who received a study vaccination and provided evaluable serum samples both at day 1 and at day 22
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | aTIV (Pooled) | Licensed TIV
Number analyzed (Participants) | 3479 | 3482
Titers
  H1N1 strain (N=3477,3480) | 196 [184 to 208] | 142 [134 to 151]
  H3N2 strain (N=3477,3479) | 534 [506 to 563] | 334 [317 to 353]
  B strain | 54 [51 to 57] | 48 [45 to 50]
Statistical Analysis 1: Comparison: aTIV (Pooled) vs Licensed TIV; Superiority was established if the lower bound of the 95% CI for the day 22 vaccine group GMT ratios for at least 2 homologous strains was >1.5; Test type: Superiority or Other; GMT ratio (H1N1 strain) = 1.37, 95% CI 2-sided [1.29 to 1.46]
Statistical Analysis 2: Comparison: aTIV (Pooled) vs Licensed TIV; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; GMT ratio (H3N2 strain) = 1.60, 95% CI 2-sided [1.51 to 1.68]
Statistical Analysis 3: Comparison: aTIV (Pooled) vs Licensed TIV; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; GMT ratio (B strain) = 1.14, 95% CI 2-sided [1.08 to 1.2]

5. Primary Outcome: Comparison of aTIV Versus TIV in Terms of Percentage of Subjects Achieving Seroconversion Against Homologous Strains-FAS
Description: The superiority of HI antibody responses of aTIV compared to TIV assessed in terms of percentage of subjects achieving seroconversion at three weeks after vaccination against the three homologous vaccine strains.
  Seroconversion defined as prevaccination HI titer <10 and postvaccination HI titer ≥40 or at least a 4-fold increase in HI titers from prevaccination HI titer ≥10.
Time Frame: Day 22 post vaccination
Population: Analysis was done on FAS.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | aTIV (Pooled) | Licensed TIV
Number analyzed (Participants) | 3479 | 3482
Percentage of subjects
  H1N1 strain (N=3477, 3480) | 77.3 [75.8 to 78.6] | 67.8 [66.2 to 69.3]
  H3N2 strain (N=3477,3479) | 73.7 [72.2 to 75.1] | 60.6 [59.0 to 62.2]
  B strain | 46.9 [45.3 to 48.6] | 41.5 [39.8 to 43.1]
Statistical Analysis 1: Comparison: aTIV (Pooled) vs Licensed TIV; Superiority was established if the lower bound of the 95% CI for the day 22 differences in seroconversion rates for at least 2 homologous strains was >10%; Test type: Superiority or Other; Group difference (H1N1 strain) = 8.9, 95% CI 2-sided [6.9 to 10.9]
Statistical Analysis 2: Comparison: aTIV (Pooled) vs Licensed TIV; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; Group difference (H3N2 strain) = 12.7, 95% CI 2-sided [10.6 to 14.8]
Statistical Analysis 3: Comparison: aTIV (Pooled) vs Licensed TIV; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; Group difference (B strain) = 5.1, 95% CI 2-sided [2.9 to 7.2]

6. Primary Outcome: Percentage of Subjects With HI Titers ≥40 Against Homologous Strains
Description: The percentage of subjects demonstrating HI titers ≥40, in overall group and in subjects with pre-defined co-morbidities (high risk group), against homologous strains, three weeks after vaccination with aTIV or TIV.
Time Frame: Day 22 post vaccination
Population: Analysis was done on the FAS.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | aTIV (Pooled) | Licensed TIV
Number analyzed (Participants) | 3479 | 3482
Percentage of subjects
  H1N1 strain (N=3477,3480) overall | 91.1 [90.1 to 92.0] | 84.5 [83.3 to 85.7]
  H3N2 strain (N=3477,3479) overall | 99.0 [98.6 to 99.3] | 97.0 [96.4 to 97.6]
  B strain, overall | 64.6 [62.9 to 66.2] | 58.9 [57.3 to 60.6]
  H1N1 strain (N=1299,1273), high risk group | 91.9 [90.3 to 93.3] | 85.8 [83.7 to 87.7]
  H3N2 strain (N=1299,1273), high risk group | 98.7 [97.9 to 99.2] | 96.7 [95.6 to 97.6]
  B strain (N=1300,1273), high risk group | 66.3 [63.7 to 68.9] | 61.4 [58.7 to 64.1]

7. Primary Outcome: Percentage of Subjects Achieving Seroconversion in HI Titers, Against Homologous Strains
Description: The percentage of subjects achieving seroconversion in HI titers from baseline, in overall group and in subjects with pre-defined co-morbidities (high risk group), against homologous strains, three weeks after vaccination with aTIV or TIV.
  Seroconversion is defined as prevaccination HI titer <10 and postvaccination HI titer ≥40 or at least a 4-fold increase in HI titers from prevaccination HI titer ≥10.
Time Frame: Day 22 post vaccination
Population: Analysis was done on the FAS.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | aTIV (Pooled) | Licensed TIV
Number analyzed (Participants) | 3479 | 3482
Percentage of subjects
  H1N1 strain ( N= 3477,3480), overall | 77.3 [75.8 to 78.6] | 67.8 [66.2 to 69.3]
  H3N2 strain ( N= 3477,3479), overall | 73.7 [72.2 to 75.1] | 60.6 [59.0 to 62.2]
  B strain, overall | 46.9 [45.3 to 48.6] | 41.5 [39.8 to 43.1]
  H1N1 strain ( N= 1299,1273), high risk group | 72.6 [70.1 to 75.0] | 62.0 [59.3 to 64.7]
  H3N2 strain ( N= 1299,1273), high risk group | 68.9 [66.3 to 71.4] | 55.2 [52.4 to 58.0]
  B strain (N= 1299,1273), high risk group | 40.0 [37.3 to 42.7] | 34.3 [31.6 to 36.9]

8. Primary Outcome: Geometric Mean Ratio (GMR) of Post- Versus Pre-vaccination HI Titers Against Homologous Strains
Description: The GMR of post-vaccination versus pre-vaccination HI titers (day 22/day 1) in overall group and in subjects with pre-defined co-morbidities (high risk group), against homologous strains, three weeks after vaccination with aTIV or TIV.
Time Frame: Day 22 post vaccination
Population: Analysis was done on the FAS
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | aTIV (Pooled) | Licensed TIV
Number analyzed (Participants) | 3479 | 3482
Ratio
  H1N1 strain (N=3477, 3480), overall | 13 [13 to 14] | 9.77 [9.14 to 10]
  H3N2 strain (N=3477, 3479), overall | 10 [9.48 to 11] | 6.54 [6.06 to 7.06]
  B strain , overall | 4.85 [4.59 to 5.13] | 4.27 [4.04 to 4.52]
  H1N1 strain (N=1299, 1273), high risk group | 12 [11 to 14] | 9.17 [8.28 to 10]
  H3N2 strain (N=1299, 1273), high risk group | 9.26 [8.31 to 10] | 6.24 [5.59 to 6.96]
  B strain (N=1300, 1273), high risk group | 4.48 [4.14 to 4.84] | 3.99 [3.68 to 4.31]

9. Secondary Outcome: Comparison of aTIV Versus TIV in High Risk Group in Terms of GMTs Against Homologous Strains-PPS
Description: The non-inferiority of HI antibody responses of ATIV compared to TIV, in subjects with pre-defined co-morbidities (high risk subjects), was assessed in terms of post vaccination GMTs at three weeks after vaccination against the three homologous vaccine strains.
Time Frame: Day 22 post vaccination
Population: Analysis was done on PPS.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | aTIV (Pooled) | Licensed TIV
Number analyzed (Participants) | 1195 | 1190
Titers
  H1N1 strain (1194, 1190) | 221 [201 to 243] | 161 [146 to 177]
  H3N2 strain (1194, 1190) | 519 [477 to 565] | 331 [304 to 360]
  B strain | 61 [56 to 66] | 54 [50 to 59]
Statistical Analysis 1: Comparison: aTIV (Pooled) vs Licensed TIV; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; GMT ratio (H1N1 strain) = 1.38, 95% CI 2-sided [1.25 to 1.52]
Statistical Analysis 2: Comparison: aTIV (Pooled) vs Licensed TIV; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; GMT ratio (H3N2 strain) = 1.57, 95% CI 2-sided [1.44 to 1.72]
Statistical Analysis 3: Comparison: aTIV (Pooled) vs Licensed TIV; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; GMT ratio (B strain) = 1.12, 95% CI 2-sided [1.03 to 1.21]

10. Secondary Outcome: Comparison of HI Antibody Responses of aTIV Versus TIV, in High Risk Group in Terms of Percentage of Subjects Achieving Seroconversion Against Homologous Strains-PPS
Description: The non-inferiority of HI antibody responses of ATIV compared to TIV, in subjects with pre-defined co-morbidities (high risk group), assessed in terms of percentage of subjects achieving seroconversion at three weeks after vaccination against the homologous vaccine strains.
  Seroconversion is defined as prevaccination HI titer <10 and postvaccination HI titer ≥40 or at least a 4-fold increase in HI titers from prevaccination HI titer ≥10.
Time Frame: Day 22 post vaccination
Population: Analysis was done on PPS.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | aTIV (Pooled) | Licensed TIV
Number analyzed (Participants) | 1195 | 1190
Percentage of subjects
  H1N1 strain (N=1194, 1190) | 73.6 [71.0 to 76.1] | 61.7 [58.9 to 64.5]
  H3N2 strain (N=1194, 1190) | 69.1 [66.4 to 71.7] | 54.8 [51.9 to 57.6]
  B strain | 40.0 [37.2 to 42.8] | 34.0 [31.3 to 36.7]
Statistical Analysis 1: Comparison: aTIV (Pooled) vs Licensed TIV; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Group difference (H1N1 strain) = 11.1, 95% CI 2-sided [7.5 to 14.6]
Statistical Analysis 2: Comparison: aTIV (Pooled) vs Licensed TIV; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Group difference (H3N2 strain) = 13.5, 95% CI 2-sided [9.8 to 17.2]
Statistical Analysis 3: Comparison: aTIV (Pooled) vs Licensed TIV; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Group difference (B strain) = 5.0, 95% CI 2-sided [1.4 to 8.5]

11. Secondary Outcome: Comparison of aTIV Versus TIV in High Risk Group in Terms of GMTs Against Homologous Strains-FAS
Description: The superiority of HI antibody responses of aTIV compared to TIV, in subjects with predefined co-morbidities (high risk group) assessed in terms of post vaccination GMTs at three weeks after vaccination against the three homologous vaccine strains.
Time Frame: Day 22 post vaccination
Population: Analysis was done on FAS population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | aTIV (Pooled) | Licensed TIV
Number analyzed (Participants) | 1300 | 1273
Titers
  H1N1 strain (N=1299,1273) | 212 [194 to 232] | 160 [147 to 176]
  H3N2 strain (N=1299,1273) | 499 [460 to 540] | 324 [299 to 351]
  B strain | 60 [55 to 64] | 54 [50 to 58]
Statistical Analysis 1: Comparison: aTIV (Pooled) vs Licensed TIV; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; GMT ratio (H1N1 strain) = 1.32, 95% CI 2-sided [1.2 to 1.45]
Statistical Analysis 2: Comparison: aTIV (Pooled) vs Licensed TIV; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; GMT ratio (H3N2 strain) = 1.54, 95% CI 2-sided [1.42 to 1.68]
Statistical Analysis 3: Comparison: aTIV (Pooled) vs Licensed TIV; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; GMT ratio (B strain) = 1.11, 95% CI 2-sided [1.03 to 1.21]

12. Primary Outcome: Percentage of Subjects With HI Titers ≥40 Against Heterologous Strains
Description: The percentage of subjects demonstrating HI titers ≥40, in overall group and in subjects with pre-defined co-morbidities (high risk group), against heterologous strains, three weeks after vaccination with aTIV or TIV.
Time Frame: Day 22 post vaccination
Population: Analysis was done on the FAS.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | aTIV (Pooled) | Licensed TIV
Number analyzed (Participants) | 887 | 881
Percentage of subjects
  H3N2/Brisbane strain(N=887,880), overall | 95.8 [94.3 to 97.1] | 94.0 [92.2 to 95.5]
  H3N2/Wisconsin strain, overall | 99.6 [98.9 to 99.9] | 98.4 [97.4 to 99.1]
  B strain (N=887,880), overall | 76.2 [73.3 to 79.0] | 72.4 [69.3 to 75.3]
  H3N2/Brisbane (N=330, 333), high risk group | 94.9 [91.9 to 97.0] | 94.0 [90.9 to 96.3]
  H3N2/Wisconsin (N=330, 333), high risk group | 99.7 [98.3 to 100] | 98.5 [96.5 to 99.5]
  B strain (N=330, 333), high risk group | 83.3 [78.9 to 87.2] | 78.4 [73.6 to 82.7]

13. Primary Outcome: Geometric Mean Ratio (GMR) of Post- Versus Pre-vaccination HI Titers, Against Heterologous Strains
Description: The GMR of post-vaccination versus pre-vaccination HI titers (day 22/day 1) in overall group and in subjects with pre-defined co-morbidities (high risk group), against heterologous strains, three weeks after vaccination with aTIV or TIV.
Time Frame: Day 22 post vaccination
Population: Analysis was done on the FAS.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | aTIV (Pooled) | Licensed TIV
Number analyzed (Participants) | 887 | 881
Ratio
  H3N2/Brisbane strain (N=887,880), overall | 5.76 [5.02 to 6.6] | 3.87 [3.37 to 4.44]
  H3N2/Wisconsin strain, overall | 4.95 [4.36 to 5.62] | 3.54 [3.12 to 4.03]
  B strain (N=887,880), overall | 5.76 [5.2 to 6.38] | 5.28 [4.76 to 5.85]
  H3N2/Brisbane strain (N=330,333), high risk group | 5.42 [4.47 to 6.57] | 4.15 [3.43 to 5.03]
  H3N2/Wisconsin strain (N=330,333), high risk group | 4.67 [3.87 to 5.62] | 3.73 [3.1 to 4.49]
  B strain (N=330,333), high risk group | 5.41 [4.66 to 6.28] | 4.77 [4.11 to 5.53]

14. Primary Outcome: Percentage of Subjects Achieving Seroconversion in HI Titers, Against Heterologous Strains
Description: The percentage of subjects achieving seroconversion in HI titers from baseline, in overall group and in subjects with pre-defined co-morbidities (high risk group), against heterologous strains, three weeks after vaccination with aTIV or TIV.
  Seroconversion is defined as prevaccination HI titer <10 and postvaccination HI titer ≥40 or at least a 4-fold increase in HI titers from prevaccination HI titer ≥10.
Time Frame: Day 22 post vaccination
Population: Analysis was done on the FAS.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | aTIV (Pooled) | Licensed TIV
Number analyzed (Participants) | 887 | 881
Percentage of subjects
  H3N2/Brisbane, overall (N=887, 880) | 60.4 [57.1 to 63.7] | 48.4 [45.1 to 51.8]
  H3N2/Wisconsin, overall | 57.5 [54.2 to 60.8] | 45.5 [42.2 to 48.9]
  B strain, overall (N=887, 880) | 53.3 [50.0 to 56.7] | 49.8 [46.4 to 53.1]
  H3N2/Brisbane (N= 330,333), high risk group | 54.2 [48.7 to 59.7] | 41.4 [36.1 to 46.9]
  H3N2/Wisconsin ( N= 330,333), high risk group | 52.1 [46.6 to 57.6] | 38.7 [33.5 to 44.2]
  B strain (N= 330, 333), high risk group | 46.4 [40.9 to 51.9] | 41.7 [36.4 to 47.2]

15. Secondary Outcome: Comparison of HI Antibody Responses of aTIV Versus TIV, in High Risk Group in Terms of Percentage of Subjects Achieving Seroconversion Against Homologous Strains-FAS
Description: The superiority of HI antibody responses of aTIV compared to TIV, in subjects with pre-defined co-morbidities (high risk group), assessed in terms of percentage of subjects achieving seroconversion at three weeks after vaccination against the homologous vaccine strains.
  Seroconversion is defined as prevaccination HI titer <10 and postvaccination HI titer ≥40 or at least a 4-fold increase in HI titers from prevaccination HI titer ≥10.
Time Frame: Day 22 postvaccination
Population: Analysis was done on FAS.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | aTIV (Pooled) | Licensed TIV
Number analyzed (Participants) | 1300 | 1273
Percentage of subjects
  H1N1 strain (N=1299,1273) | 72.6 [70.1 to 75.0] | 62.0 [59.3 to 64.7]
  H3N2 strain (N=1299,1273) | 68.9 [66.3 to 71.4] | 55.2 [52.4 to 58.0]
  B strain | 40.0 [37.3 to 42.7] | 34.3 [31.6 to 36.9]
Statistical Analysis 1: Comparison: aTIV (Pooled) vs Licensed TIV; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; Group difference (H1N1 strain) = 9.9, 95% CI 2-sided [6.4 to 13.3]
Statistical Analysis 2: Comparison: aTIV (Pooled) vs Licensed TIV; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; Group difference (H3N2 strain) = 13.0, 95% CI 2-sided [9.5 to 16.6]
Statistical Analysis 3: Comparison: aTIV (Pooled) vs Licensed TIV; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; Group difference (B strain) = 4.9, 95% CI 2-sided [1.5 to 8.3]

16. Secondary Outcome: Comparison of aTIV Versus TIV in Terms of GMTs Against Heterologous Strains-PPS
Description: The non-inferiority of HI antibody responses of aTIV compared to TIV against the heterologous vaccine strains, in overall group and in subjects with pre-defined co-morbidities (high risk subjects), was assessed in terms of post vaccination GMTs at three weeks after vaccination .
Time Frame: Day 22 post vaccination
Population: Analysis was done on PPS.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | aTIV (Pooled) | Licensed TIV
Number analyzed (Participants) | 834 | 815
Titers
  H3N2/Brisbane (overall) (N=834,814) | 369 [329 to 414] | 255 [227 to 287]
  H3N2/Wisconsin (overall) | 1037 [940 to 1144] | 764 [691 to 846]
  B strain (overall) (N=834,814) | 89 [80 to 99] | 82 [73 to 91]
  H3N2/Brisbane (high risk) (N=302,307) | 377 [319 to 445] | 279 [236 to 330]
  H3N2/Wisconsin (high risk) (N=302,307) | 965 [831 to 1121] | 751 [646 to 873]
  B strain (high risk) (N=302,307) | 117 [100 to 136] | 105 [90 to 123]
Statistical Analysis 1: Comparison: aTIV (Pooled) vs Licensed TIV; Test type: Non-Inferiority or Equivalence — Non-inferiority was established if the lower bound of the 95% CI for the day 22 vaccine group GMT ratios for all 3 heterologous strains was >0.67; GMT Ratio (H3N2/Brisbane-overall) = 1.45, 95% CI 2-sided [1.29 to 1.63]
Statistical Analysis 2: Comparison: aTIV (Pooled) vs Licensed TIV; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 16, analysis 1]; GMT Ratio (H3N2/Wisconsin-overall) = 1.36, 95% CI 2-sided [1.23 to 1.5]
Statistical Analysis 3: Comparison: aTIV (Pooled) vs Licensed TIV; Test type: Non-Inferiority or Equivalence — Non-inferiority was established if the lower bound of the 95% CI for the day 22 vaccine group GMT ratios for all 3 heterologous strains was ≥0.67; GMT Ratio (B strain-overall) = 1.09, 95% CI 2-sided [0.98 to 1.21]
Statistical Analysis 4: Comparison: aTIV (Pooled) vs Licensed TIV; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 16, analysis 1]; GMT Ratio(H3N2/Brisbane-high risk group) = 1.35, 95% CI [1.13 to 1.61]
Statistical Analysis 5: Comparison: aTIV (Pooled) vs Licensed TIV; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 16, analysis 1]; GMT Ratio(H3N2/Wisconsin-high risk group = 1.29, 95% CI 2-sided [1.1 to 1.5]
Statistical Analysis 6: Comparison: aTIV (Pooled) vs Licensed TIV; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 16, analysis 1]; GMT Ratio (B strain-high risk group) = 1.11, 95% CI 2-sided [0.95 to 1.3]

17. Secondary Outcome: Comparison of aTIV Versus TIV in Terms of GMTs Against Heterologous Strains-FAS
Description: The superiority of HI antibody responses of aTIV compared to TIV against the heterologous vaccine strains, in overall group and in subjects with pre-defined co-morbidities (high risk subjects), was assessed in terms of post vaccination GMTs at three weeks after vaccination.
Time Frame: Day 22 post vaccination
Population: Analysis was done on FAS.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | aTIV (Pooled) | Licensed TIV
Number analyzed (Participants) | 887 | 881
Titers
  H3N2/Brisbane (overall) (N=887,880) | 362 [325 to 404] | 243 [218 to 271]
  H3N2/Wisconsin (overall) | 1016 [926 to 1115] | 738 [672 to 811]
  B strain (overall) (N=887,880) | 87 [79 to 97] | 80 [72 to 88]
  H3N2/Brisbane (high risk) (N=302,307) | 364 [312 to 425] | 267 [229 to 312]
  H3N2/Wisconsin (high risk) (N=302,307) | 927 [807 to 1065] | 724 [631 to 831]
  B strain (high risk) (N=302,307) | 112 [97 to 129] | 99 [87 to 114]
Statistical Analysis 1: Comparison: aTIV (Pooled) vs Licensed TIV; Superiority was established if the lower bound of the 95% CI for the day 22 vaccine group GMT ratios for at least 2 heterologous strains was >1.5; Test type: Superiority or Other; GMT ratio (H3N2/Brisbane-overall) = 1.49, 95% CI 2-sided [1.33 to 1.67]
Statistical Analysis 2: Comparison: aTIV (Pooled) vs Licensed TIV; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; GMT ratio(H3N2/Wisconsin-overall) = 1.38, 95% CI 2-sided [1.25 to 1.52]
Statistical Analysis 3: Comparison: aTIV (Pooled) vs Licensed TIV; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; GMT ratio (B strain-overall) = 1.09, 95% CI 2-sided [0.99 to 1.21]
Statistical Analysis 4: Comparison: aTIV (Pooled) vs Licensed TIV; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; GMT ratio (H3N2/Brisbane-high risk) = 1.36, 95% CI 2-sided [1.15 to 1.61]
Statistical Analysis 5: Comparison: aTIV (Pooled) vs Licensed TIV; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; GMT ratio(H3N2/Wisconsin-high risk) = 1.28, 95% CI 2-sided [1.1 to 1.48]
Statistical Analysis 6: Comparison: aTIV (Pooled) vs Licensed TIV; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; GMT ratio (B strain-high risk) = 1.13, 95% CI 2-sided [0.97 to 1.31]

18. Secondary Outcome: Comparison of HI Antibody Responses of aTIV Versus TIV, in Terms of Percentage of Subjects Achieving Seroconversion Against Heterologous Strains-PPS
Description: The non-inferiority of HI antibody responses of aTIV compared to TIV against the heterologous strains, in overall group and in subjects with pre-defined co-morbidities (high risk group), assessed in terms of percentage of subjects achieving seroconversion at three weeks after vaccination.
  Seroconversion is defined as prevaccination HI titer <10 and postvaccination HI titer ≥40 or at least a 4-fold increase in HI titers from prevaccination HI titer ≥10.
Time Frame: Day 22 postvaccination
Population: Analysis was done on PPS.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | aTIV (Pooled) | Licensed TIV
Number analyzed (Participants) | 834 | 815
Percentage of subjects
  H3N2/Brisbane (overall) (N=834,814) | 60.0 [56.5 to 63.3] | 49.1 [45.7 to 52.6]
  H3N2/Wisconsin (overall) | 57.0 [53.5 to 60.4] | 45.9 [42.4 to 49.4]
  B strain (overall) (N=834,814) | 52.8 [49.3 to 56.2] | 49.3 [45.8 to 52.8]
  H3N2/Brisbane (high risk) (N=302,307) | 54.3 [48.5 to 60.0] | 41.7 [36.1 to 47.4]
  H3N2/Wisconsin (high risk) (N=302,307) | 51.7 [45.9 to 57.4] | 38.8 [33.3 to 44.5]
  B strain (high risk) (N=302,307) | 45.7 [40.0 to 51.5] | 41.4 [35.8 to 47.1]
Statistical Analysis 1: Comparison: aTIV (Pooled) vs Licensed TIV; Test type: Non-Inferiority or Equivalence — Non-inferiority was established if the lower bound of the 95% CI for the day 22 differences in seroconversion rates for all 3 heterologous strains was ≥-10%; Group difference (H3N2/Brisbane-overall) = 11.3, 95% CI 2-sided [6.7 to 15.9]
Statistical Analysis 2: Comparison: aTIV (Pooled) vs Licensed TIV; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 18, analysis 1]; Group difference(H3N2/Wisconsin-overall) = 11.9, 95% CI 2-sided [7.3 to 16.6]
Statistical Analysis 3: Comparison: aTIV (Pooled) vs Licensed TIV; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Slope = 4.0, 95% CI 2-sided [-0.4 to 8.4]
Statistical Analysis 4: Comparison: aTIV (Pooled) vs Licensed TIV; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 18, analysis 1]; Group difference(H3N2/Brisbane-high risk = 12.3, 95% CI 2-sided [4.8 to 19.9]
Statistical Analysis 5: Comparison: aTIV (Pooled) vs Licensed TIV; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Group difference(H3N2Wisconsin-high risk = 12.6, 95% CI 2-sided [5.0 to 20.2]
Statistical Analysis 6: Comparison: aTIV (Pooled) vs Licensed TIV; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 18, analysis 1]; Group difference (B strain-high risk) = 4.8, 95% CI 2-sided [-2.1 to 11.8]

19. Secondary Outcome: Comparison of aTIV Versus TIV in Terms of Percentage of Subjects Achieving Seroconversion Against Heterologous Strains-FAS
Description: The superiority of HI antibody responses of aTIV compared to TIV against the heterologous vaccine strains, in overall group and in subjects with pre-defined co-morbidities (high risk subjects), was assessed in terms of percentage of subjects achieving seroconversion, at three weeks after vaccination.
  Seroconversion is defined as prevaccination HI titer <10 and postvaccination HI titer ≥40 or at least a 4-fold increase in HI titers from prevaccination HI titer ≥10.
Time Frame: Day 22 post vaccination
Population: Analysis was done on FAS
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | aTIV (Pooled) | Licensed TIV
Number analyzed (Participants) | 887 | 881
Percentage of subjects
  H3N2/Brisbane (overall) (N=887,880) | 60.4 [57.1 to 63.7] | 48.4 [45.1 to 51.8]
  H3N2/Wisconsin (overall) | 57.5 [54.2 to 60.8] | 45.5 [42.2 to 48.9]
  B strain (overall) (N=887,880) | 53.3 [50.0 to 56.7] | 49.8 [46.4 to 53.1]
  H3N2/Brisbane (high risk) (N=330, 333) | 54.2 [48.7 to 59.7] | 41.4 [36.1 to 46.9]
  H3N2/Wisconsin (high risk) (N=330,333) | 52.1 [46.6 to 57.6] | 38.7 [33.5 to 44.2]
  B strain (high risk) (N=330, 333) | 46.4 [40.9 to 51.9] | 41.7 [36.4 to 47.2]
Statistical Analysis 1: Comparison: aTIV (Pooled) vs Licensed TIV; Superiority was established if the lower bound of the 95% CI for the day 22 differences in seroconversion rates for at least 2 heterologous strains was >10%; Test type: Superiority or Other; Group difference (H3N2/Brisbane-overall) = 12.5, 95% CI 2-sided [8.1 to 16.9]
Statistical Analysis 2: Comparison: aTIV (Pooled) vs Licensed TIV; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; Group difference(H3N2/Wisconsin-overall) = 12.6, 95% CI 2-sided [8.1 to 17.1]
Statistical Analysis 3: Comparison: aTIV (Pooled) vs Licensed TIV; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; Group difference (B strain-overall) = 4.6, 95% CI 2-sided [0.4 to 8.8]
Statistical Analysis 4: Comparison: aTIV (Pooled) vs Licensed TIV; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; Group difference(H3N2/Brisbane-high risk = 12.4, 95% CI 2-sided [5.2 to 19.6]
Statistical Analysis 5: Comparison: aTIV (Pooled) vs Licensed TIV; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; Group difference(H3N2/Wisconsin-highrisk = 13.0, 95% CI 2-sided [5.8 to 20.3]
Statistical Analysis 6: Comparison: aTIV (Pooled) vs Licensed TIV; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; Group difference (B strain-high risk) = 5.1, 95% CI 2-sided [-1.6 to 11.8]

20. Secondary Outcome: Persistence of GMTs Against Homologous and Heterologous Strains
Description: The GMTs against homologous and heterologous strains, persisting in subjects at six months (day 181) and one year (day 366) after vaccination with either aTIV or TIV.
Time Frame: Day 181, Day 366 post vaccination
Population: The analysis was done on the FAS (persistence) subset population i.e all randomized population only from US sites who received a study vaccination, provided evaluable blood samples at day 1, day 22, day 181, and day 366.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | aTIV (Pooled) | Licensed TIV
Number analyzed (Participants) | 189 | 191
Titers
  H1N1 (homologous) Day 181 | 71 [60 to 84] | 68 [57 to 80]
  H1N1 (homologous) Day 366 | 49 [41 to 59] | 52 [44 to 63]
  H3N2 (homologous) Day 181 | 123 [104 to 146] | 91 [77 to 108]
  H3N2 (homologous) Day 366 | 70 [59 to 84] | 54 [45 to 64]
  B (homologous) Day 181 | 25 [21 to 29] | 22 [19 to 26]
  B (homologous) Day 366 | 21 [18 to 24] | 20 [17 to 23]
  B (heterologous) Day 181 | 39 [33 to 45] | 38 [33 to 44]
  B (heterologous) Day 366 | 38 [33 to 44] | 40 [35 to 46]
  H3N2/Brisbane (heterologous) Day 181 | 100 [84 to 120] | 81 [68 to 97]
  H3N2/Brisbane(heterologous) Day 366 | 75 [63 to 90] | 72 [60 to 86]
  H3N2/Wisconsin (heterologous) Day 181 | 228 [189 to 275] | 194 [161 to 233]
  H3N2/Wisconsin (heterologous) Day 366 | 190 [157 to 231] | 182 [150 to 221]

21. Secondary Outcome: Percentage of Subjects With Seroconversion Upto One Year After Vaccination, Against Homologous and Heterologous Strains
Description: The percentage of subjects demonstrating seroconversion in HI titers against homologous and heterologous strains, at six months (day 181) and one year (day 366) after vaccination with either aTIV or TIV.
  Seroconversion is defined as prevaccination HI titer <10 and postvaccination HI titer ≥40 or at least a 4-fold increase in HI titers from prevaccination HI titer ≥10.
Time Frame: Day 181, Day 366 post vaccination
Population: The analysis was done on the FAS (persistence) subset.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | aTIV (Pooled) | Licensed TIV
Number analyzed (Participants) | 189 | 191
Percentage of subjects
  H1N1 (homologous) Day 181 | 28.6 [22.3 to 35.6] | 26.2 [20.1 to 33]
  H1N1 (homologous) Day 366 | 18.5 [13.3 to 24.8] | 19.4 [14.0 to 25.7]
  H3N2 (homologous) Day 181 | 36.0 [29.1 to 43.3] | 24.6 [18.7 to 31.4]
  H3N2 (homologous) Day 366 | 16.9 [11.9 to 23.1] | 12.6 [8.2 to 18.1]
  B (homologous) Day 181 | 3.7 [1.5 to 7.5] | 2.6 [0.9 to 6.0]
  B (homologous) Day 366 | 2.1 [0.6 to 5.3] | 3.1 [1.2 to 6.7]
  B (heterologous) Day 181 | 2.65 [0.86 to 6.07] | 3.14 [1.16 to 6.71]
  B (heterologous) Day 366 | 4.23 [1.84 to 8.17] | 3.14 [1.16 to 6.71]
  H3N2/Brisbane (heterologous) Day 181 | 15.34 [10.52 to 21.29] | 8.38 [4.86 to 13.25]
  H3N2/Brisbane(heterologous) Day 366 | 7.94 [4.51 to 12.75] | 5.24 [2.54 to 9.42]
  H3N2/Wisconsin (heterologous) Day 181 | 12.17 [7.87 to 17.70] | 8.90 [5.27 to 13.87]
  H3N2/Wisconsin (heterologous) Day 366 | 8.99 [5.33 to 14.01] | 6.28 [3.29 to 10.72]

22. Secondary Outcome: Number of Subjects Reporting Influenza Like Illness (ILI) Across Vaccine Groups
Description: The number of subjects reporting ILI from three weeks after vaccination to up to one year in aTIV group compared to TIV group, by country.
Time Frame: Day 22 through Day 366 post vaccination
Population: Analysis was done on the modified full analysis set (mFAS; effectiveness) population i.e all subjects in the randomized population who received a study vaccination but excluding those who received a non-study vaccine during the follow-up phase.
Measure: Number; unit: participants
Arm/Group | aTIV (Pooled) | Licensed TIV
Number analyzed (Participants) | 3497 | 3498
participants
  Columbia (N=516, 506) | 119 | 97
  Panama (N=108, 102) | 20 | 21
  Philippines (N=1836,1835) | 102 | 113
  United states (N=1037,1055) | 72 | 76

23. Secondary Outcome: Number of High Risk Subjects With Exacerbation of Preexisting Chronic Disease, Across Vaccine Groups
Description: The number of high risk subjects reporting exacerbation of preexisting chronic conditions (i.e.congestive heart failure, Chronic Obstructive Pulmonary disease (COPD), asthma, hepatic disease, renal insufficiency, and neurological/neuromuscular or metabolic disorders including diabetes mellitus) in aTIV group compared to TIV group.
Time Frame: Day 1 through Day 366 post vaccination
Population: Analysis was done on the mFAS (effectiveness) population.
Measure: Number; unit: participants
Arm/Group | aTIV (Pooled) | Licensed TIV
Number analyzed (Participants) | 1307 | 1281
participants | 55 | 48

24. Secondary Outcome: Number of Subjects Reporting Healthcare Utilization Across Vaccine Groups
Description: The number of subjects with emergency room visits, unscheduled physician visits, and hospitalizations due to community acquired influenza or pneumonia, cardiopulmonary disease, cardiac disease, respiratory or pulmonary disease,in aTIV group compared to TIV group.
Time Frame: Day 1 through Day 366 post vaccination
Population: Analysis was done on the mFAS (effectiveness).
Measure: Number; unit: participants
Arm/Group | aTIV (Pooled) | Licensed TIV
Number analyzed (Participants) | 3499 | 3502
participants | 275 | 289

25. Secondary Outcome: All Cause Mortality Rate, Across Vaccine Groups
Description: The all-cause mortality rate (excluding injury)reported in aTIV group compared to TIV group, by country.
Time Frame: Day 1 through Day 366 post vaccination
Population: Analysis was done on the mFAS (effectiveness).
Measure: Number; unit: participants
Arm/Group | aTIV (Pooled) | Licensed TIV
Number analyzed (Participants) | 3540 | 3541
participants
  Columbia (N=519, 509) | 7 | 7
  Panama (N=109, 105) | 0 | 0
  Philippines (N=1873,1867) | 39 | 34
  United states (N=1039,1060) | 6 | 5

26. Secondary Outcome: Number of Subjects Reporting Solicited Adverse Events Following Vaccination
Description: The number of subjects reporting solicited local and systemic adverse events and other adverse events in aTIV group compared to TIV group.
Time Frame: Day 1 through Day 7 post vaccination
Population: Analysis was done on the safety set i.e all randomized subjects who received a study vaccination and provided postvaccination safety data.
Measure: Number; unit: participants
Arm/Group | aTIV (Pooled) | Licensed TIV
Number analyzed (Participants) | 3505 | 3495
participants
  Any Local | 1137 | 593
  Injection site erythema (N=3492, 3485) | 43 | 18
  Injection site induration (N=3494, 3488) | 45 | 17
  Injection site tenderness (N=3495,3483) | 739 | 391
  Injection site swelling (N=3495,3488) | 43 | 15
  Injection site pain (N=3495,3485) | 875 | 425
  Any sytemic | 1120 | 902
  Chills (N=3495,3485) | 235 | 163
  Myalgia (N=3496,3487) | 515 | 339
  Arthralgia (N=3492,3486) | 296 | 272
  Headache (N= 3495,3486) | 463 | 391
  Fatigue (N= 3494, 3484) | 466 | 361
  Nausea (N=3492,3482) | 101 | 98
  Vomiting (N=3494,3483) | 48 | 59
  Diarrhea (N=3494,3485) | 168 | 158
  Fever (≥ 38°C) | 122 | 116
  Any other | 210 | 165
  Oral Temperature (≥ 40°C) | 3 | 0
  Analgesic/Antipyretic used | 158 | 122

ADVERSE EVENTS:
Time Frame: Solicited adverse events (AEs) were collected from Day 1 to 7 postvaccination; unsolicited AEs from Day 1 to Day 22; Serious AEs from Day 1 to Day 366.
Arm/Group | aTIV (Pooled) | Licensed TIV
Serious Adverse Events (participants affected / at risk) | 264/3545 | 243/3537
Other Adverse Events (participants affected / at risk) | 1678/3545 | 1257/3537
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | aTIV (Pooled) (N=3545) | Licensed TIV (N=3537)
Anemia (Blood and lymphatic system disorders) | 2 | 5
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Idiopathic Thrombocytopenic coagulation (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Sideroblastic anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 2 | 0
Acute myocardial infarction (Cardiac disorders) | 11 | 7
Angina pectoris (Cardiac disorders) | 1 | 2
Angina unstable (Cardiac disorders) | 3 | 1
Arrhythmia (Cardiac disorders) | 0 | 2
Arteriosclerosis coronary artery (Cardiac disorders) | 2 | 0
Atrial Fibrillation (Cardiac disorders) | 4 | 8
Atrial tachycardia (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 2 | 0
Cardiac arrest (Cardiac disorders) | 0 | 2
Cardiac disorder (Cardiac disorders) | 2 | 0
Cardiac failure (Cardiac disorders) | 3 | 4
Cardiac failure congestive (Cardiac disorders) | 8 | 16
Cardio-respiratory arrest (Cardiac disorders) | 3 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 7 | 6
Dressler's syndrome (Cardiac disorders) | 1 | 0
Hypertensive heart disease (Cardiac disorders) | 2 | 1
Hypertrophic cardiomyopathy (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 10 | 9
Myocardial Ischemia (Cardiac disorders) | 3 | 2
Nodal arrythmia (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0
Sinus Tachycardia (Cardiac disorders) | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 2 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 1
Hydrocele (Congenital, familial and genetic disorders) | 1 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 1
Vertigo positional (Ear and labyrinth disorders) | 2 | 1
Blindness unilateral (Eye disorders) | 0 | 1
Corneal degeneration (Eye disorders) | 0 | 1
Retinal neovascularisation (Eye disorders) | 0 | 1
Viterous hemorrhage (Eye disorders) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Abdominal wall hematoma (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 0 | 1
Diverticulum (Gastrointestinal disorders) | 1 | 2
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Erosive oesophagitis (Gastrointestinal disorders) | 1 | 0
Femoral hernia,obstructive (Gastrointestinal disorders) | 1 | 0
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1
Hiatus hernia (Gastrointestinal disorders) | 1 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Ileus paralytic (Gastrointestinal disorders) | 0 | 1
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Pancreatic mass (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 4 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1
Peptic ulcer (Gastrointestinal disorders) | 0 | 4
Peptic ulcer perforation (Gastrointestinal disorders) | 1 | 0
Pneumoperitonium (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 4
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 | 7
Volvulus (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 7 | 3
Hernia obstructive (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 3 | 1
Non-cardiac chest pain (General disorders) | 1 | 1
Pyrexia (General disorders) | 1 | 2
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 7 | 2
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 4 | 4
Chronic hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 2
Arthritis bacterial (Infections and infestations) | 0 | 1
Arthritis infective (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 5 | 1
Cellulitis (Infections and infestations) | 2 | 3
Cellulitis staphylococcal (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 2
Escherichia sepsis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 5 | 6
Gastroenteritis viral (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Incision site infection (Infections and infestations) | 0 | 1
Infected skin ulcer (Infections and infestations) | 1 | 0
Infectious peritonitis (Infections and infestations) | 1 | 1
Laryngitis (Infections and infestations) | 1 | 0
Leptospirosis (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 2 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Meningitis aseptic (Infections and infestations) | 0 | 1
Peritonsillar abscess (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 32 | 35
Pneumonia viral (Infections and infestations) | 1 | 0
Pulmonary Tuberculosis (Infections and infestations) | 2 | 2
Pyelonephritis acute (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 3 | 2
Septic shock (Infections and infestations) | 3 | 3
Staphylococcal infection (Infections and infestations) | 0 | 1
Streptococcal sepsis (Infections and infestations) | 1 | 1
Tetanus (Infections and infestations) | 0 | 1
Tracheobronchitis (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 8 | 6
Urosepsis (Infections and infestations) | 0 | 1
Wound abscess (Infections and infestations) | 0 | 1
Back injury (Injury, poisoning and procedural complications) | 1 | 0
Brain herniation (Injury, poisoning and procedural complications) | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 | 1
Femur fracture (Injury, poisoning and procedural complications) | 3 | 4
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Forearm Fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 3
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0
Nerve injury (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Perirenal haematoma (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Postoperative adhesion (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal cord injury (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Traumatic liver injury (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 5 | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 | 2
Diabetic foot (Metabolism and nutrition disorders) | 2 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 0
Arthropathy (Metabolism and nutrition disorders) | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 3
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7 | 12
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder adenocarcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrointestinal stromal tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian cancer (Nervous system disorders) | 0 | 1
Pancreatic carcinoma (Nervous system disorders) | 0 | 1
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Prolymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostrate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Carotid artery disease (Nervous system disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 1
Cerebellar infraction (Nervous system disorders) | 1 | 1
Cerebral haemorrhage (Nervous system disorders) | 3 | 2
Cerebral infraction (Nervous system disorders) | 3 | 2
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 4 | 10
Cerebrovascular disorder (Nervous system disorders) | 8 | 3
Cervical myelopathy (Nervous system disorders) | 0 | 1
Cervicobrachial syndrome (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 2 | 0
Dementia alzheimer's type (Nervous system disorders) | 1 | 1
Dementia with lewy bodies (Nervous system disorders) | 1 | 0
Embolic stroke (Nervous system disorders) | 0 | 1
Guillain-barre syndrome (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 1
Headcahe (Nervous system disorders) | 0 | 1
Hemiplegia (Nervous system disorders) | 1 | 0
Ishaemic stroke (Nervous system disorders) | 0 | 3
Metabolic encephalopathy (Nervous system disorders) | 0 | 1
Radiculopathy (Nervous system disorders) | 1 | 0
Ruptured cerebral aneurysm (Nervous system disorders) | 1 | 0
Stroke in evolution (Nervous system disorders) | 0 | 1
Subarachnoid hemorrhage (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 4 | 4
Transient ischemic attack (Nervous system disorders) | 3 | 2
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 1
VIIth nerve paralysis (Nervous system disorders) | 1 | 0
Confusional state (Nervous system disorders) | 0 | 1
Mental status change (Psychiatric disorders) | 1 | 0
Azotemia (Renal and urinary disorders) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Nephropathy (Renal and urinary disorders) | 1 | 0
Obstructive uropathy (Renal and urinary disorders) | 1 | 0
Renal Failure (Renal and urinary disorders) | 2 | 0
Renal Failure acute (Renal and urinary disorders) | 3 | 2
Renal failure chronic (Renal and urinary disorders) | 2 | 2
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Endometriosis (Reproductive system and breast disorders) | 1 | 0
Prostatomegaly (Reproductive system and breast disorders) | 0 | 1
Uterovaginal prolapse (Reproductive system and breast disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 10 | 14
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angioedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aneurysm ruptured (Vascular disorders) | 0 | 1
Aortic aneurysm (Vascular disorders) | 3 | 1
Aortic dissection (Vascular disorders) | 0 | 1
Aortic stenosis (Vascular disorders) | 0 | 1
Arteriosclerosis (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 8 | 8
Hypertensive crisis (Vascular disorders) | 4 | 2
Hypotension (Vascular disorders) | 2 | 1
Peripheral artery aneurysm (Vascular disorders) | 1 | 1
Varicose ulceration (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | aTIV (Pooled) (N=3545) | Licensed TIV (N=3537)
Chills (General disorders) | 258 | 176
Fatigue (General disorders) | 480 | 379
Injection site erythema (General disorders) | 292 | 255
Injection site pain (General disorders) | 1172 | 643
Arthralgia (Musculoskeletal and connective tissue disorders) | 315 | 293
Myalgia (Musculoskeletal and connective tissue disorders) | 536 | 360
Headache (Nervous system disorders) | 492 | 426
Diarrhoea (Gastrointestinal disorders) | 186 | 172

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days